CLINICAL TRIAL: NCT03425773
Title: Single Center, Open-label, Accelerated Titration, Multiple Dosing Study to Evaluate the Safety, Tolerability, Immune Response and Pre-efficacy of BVAC-B in Patients With Progressive or Recurrent HER2/Neu Positive Gastric Cancer After Failure to Standard Care
Brief Title: Safety and Tolerability Evaluation Study of BVAC-B in Patients With HER2/Neu(Human Epithelial Growth Factor Receptor 2) Positive Gastric Cancer After Failure to Standard Care
Acronym: BVAC-B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cellid Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BVAC-B-P1
Record Dates: First submitted 2018-01-29; First posted 2018-02-08 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Stomach Neoplasms
Keywords: HER2/neu; IHC 1+; BVAC; Cellid; B-cell; Monocyte; Immunotherapeutic vaccine; Breast cancer; Colorectal cancer; Pancreatic cancer
MeSH Terms: conditions — Stomach Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Accelerated titration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BVAC-B (Experimental): BVAC-B IV injection at 0, 4, 8, 12nd weeks.
  Interventions: Biological: BVAC-B

INTERVENTIONS:
Biological: BVAC-B — Autologous B cell and monocyte presenting HER2/neu antigen

SUMMARY:
BVAC-B is immunotherapeutic vaccine using B-Cell and Monocytes as antigen presenting cell. This study is Open-label, Accelerated titration, Multiple dosing study to evaluate the safety, tolerability, immune response and pre-efficacy of BVAC-B in patients with progressive or recurrent HER2/neu positive gastric cancer after failure to standard care. 9-27 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Progressive or recurrent HER2/neu positive(IHC 1+≥) gastric cancer
* Received 1 or more chemotherapy or radiotherapy as prior therapy for progressive or recurrent tumor lesion
* At least 1 measurable lesion according to RECIST(ver 1.1)
* Ages above 19
* ECOG performance status between 0 to 2
* Patients meets the blood test standards in the screening test
* Patients meets the blood chemistry test standards in the screening test
* Patients who has agreed to a medically accepted contraceptive in this clinical trial
* Patients at least six months or more of survival can be expected
* Patients decided to participate in this clinical trial and signed written informed consent

Exclusion Criteria:

* Histopathology is a neuroendocrine or small cell carcinoma
* History of brain metastasis or signs of brain metastasis
* Clinical diagnosis of hepatitis C or hepatitis B
* Clinical diagnosis of human immunodeficiency virus (HIV)
* History of HIV infection
* Patients with heart failure, coronary artery disease(CAD) or Myocardial infarction in 6 month prior to screening. (LVEF is lower than 50% in screening visit)
* Administered the drug for other clinical trials within 4weeks before participate in this trial
* Administered any vaccines within 4weeks before participate in this trial (4 weeks for live vaccine, 2 weeks for other inactivated vaccine)
* Administered the granulocytes concentrates within 3 months before the screening visit
* Received chemotherapy or radiation therapy within 2 weeks before the 1st administration of investigational drug(BVAC-B)
* Received following formulation within 1 months before the screening visit : Chronic steroids(more than 5 days), immunosuppressant or immunomodulatory agents. G-CSF
* Patients who have participated in the clinical trial of a immunotherapeutic vaccine within 1 year or immunotherapy within 3 months before the screening visit
* Patients who is pregnant or breast-feeding
* Patients who researchers has determined that participation in the clinical trial is inappropriate
* Suspected to have other progressive cancer or malignant tumor needs treatment in 3 years. Completely treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, thyroid carcinoma, cervical intraepithelial neoplasia are not included

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
Evaluate Maximum tolerated dose(MTD) for phase 2 trial | End of Dose-escalation stage(7 month from study start, Estimated)
  Find Serious adverse drug reaction(Grade 3)
Incidence of Serious Adverse Events assessed with CTCAE v4.03 | 14th week from first injection
  Evaluate safety and tolerability

SECONDARY OUTCOMES:
Serum cytokine | Screening visit, Visit 2 (0 week) , visit 4 (4 week) ,visit 5 (6 week), visit 6 (8 week), visit 8(12 week), Termination visit(16 week)
  Measure Interferon(IFN)-r, Interleukin(IL)-4
HER2/neu specific antibody | Screening visit, every 2 weeks after 1st injection(till 16th week)
  Measure HER2/neu specific antibody concentration
NKT/NK cell assay | Screening visit, every 24hr after injection(up to 12th week)
  Measure NKT/NK cell activity
CD4/CD8 assay | Screening visit, every 2 weeks after 1st injection(up to 16th week)
  Measure CD4/CD8 T cell activity
Lymphocyte subset | Screening visit, visit 4 (4 week), visit 6 (8 week), visit 8 (12 week), termination visit (16 week)
  Measure change of lymphocyte subset
Change of tumor burden | Screening visit, Termination visit(16th week)
  Measure change of tumor burden by CT/MRI to determine pre-effecacy

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seodaemun-gu, South Korea